CLINICAL TRIAL: NCT02184910
Title: Usefulness of Serum Pepsinogen and Gastrin as the Predictive Biomarker of Atrophic Gastritis, Intestinal Metaplasia and Gastric Cancer in Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0722
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Atrophic Gastritis
Keywords: atrophic gastritis, pepsinogen, Helicobacter pylori
MeSH Terms: conditions — Gastritis, Atrophic | interventions — Pepsinogen A; Gastrins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gastritis and pepsinogen
  Interventions: Drug: pepsinogen and gastrin

INTERVENTIONS:
Drug: pepsinogen and gastrin

SUMMARY:
It is well-known that atrophic gastritis is a major risk factor for gastric cancer, which leads to variations in the serum levels of gastrin, pepsinogen (PG) I, and PGII. We want to assess the effects of age, sex, and Helicobacter pylori status on pepsinogen (PG) level for atrophic gastritis and whether gastric atrophy based on the PG test would be improved after H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

1. over 19 years
2. the patients who have gastrointestinal discomfort or get esophagogastroduodenoscopy (EGD) for health check up
3. the patients who got the procedure, endoscopic submucosal resection (ESD) for early gastric cancer

Exclusion Criteria:

1. gastrectomy history
2. advanced gastric cancer (impossible to get the gastrectomy)
3. Helicobacter eradication history
4. the patients who have chronic disease
5. cancer patients except gastric cancer within 6 months
6. who cannot perform this study according to research's decision
7. who have bleeding tendency (ex. taking antiplatelet agent, low platelet count or abnormal coagulation time)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 19 years, the patients who have gastrointestinal discomfort or get esophagastroduodenoscopy (EGD) for health check up, the patients who got the procedure, endoscopic submucosal resection (ESD) for early gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the change of pepsinogen level before and after H. pylori eradication | baseline and 6 months
  to compare the change of the pepsinogen level before and after H. pylori eradication and evaluate the correlation between the pepsinogen level and the atrophic gastritis

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea